CLINICAL TRIAL: NCT00620763
Title: Calcium Retention in Postmenopausal Women as Influenced by Beef and Other Dietary Components That Induce an Acid Load
Brief Title: Calcium Retention as Influenced by Dietary Components That Induce an Acid Load
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: USDA Grand Forks Human Nutrition Research Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: GFHNRC087; IRB-2000707-013
Record Dates: First submitted 2008-01-18; First posted 2008-02-21 (Estimated); Results first posted 2009-08-03 (Estimated); Last update posted 2018-07-02 (Actual); Status verified 2018-05

CONDITIONS: Healthy
Keywords: Meat protein; acid load; calcium retention; postmenopausal women
MeSH Terms: interventions — Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Dietary Intervention: High meat and high acid load diet followed by low meat and low acid load diet
  Interventions: Other: High Meat - High Potential Renal Acid Load (PRAL) diet; Other: Low Protein - Low Potential Renal Acid Load (PRAL) diet
- B (Experimental): Dietary Intervention: Low meat and low acid load diet followed by high meat and high acid load diet
  Interventions: Other: High Meat - High Potential Renal Acid Load (PRAL) diet; Other: Low Protein - Low Potential Renal Acid Load (PRAL) diet

INTERVENTIONS:
Other: High Meat - High Potential Renal Acid Load (PRAL) diet — Menu high in meat protein
Other: Low Protein - Low Potential Renal Acid Load (PRAL) diet — Menu low in meat protein

SUMMARY:
The impact of protein sources such as beef as part of Western diet on calcium retention remains controversial. We propose to test the hypothesis that the positive effect of high protein intake (especially from meat protein) can offset the negative effect of protein-induced net acid load on bone metabolism and the retention of body calcium. Healthy postmenopausal women recruited from the community will consume two diets differing in meat protein and acid load for 7 weeks. Calcium retention from diets will be determined using a highly sensitive measurement of whole body retention of a calcium isotope added to the diet.

ELIGIBILITY:
Inclusion Criteria:

* Average body mass index
* Normal blood work
* Normal bone density

Exclusion Criteria:

* Chronic disorder
* Non-traumatic bone fractures

Ages: 40 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2008-01; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jay Cao, PhD, Principal Investigator — USDA Grand Forks Human Nutrition Research Center
Locations (1):
- United States Department of Agriculture (USDA) Grand Forks Human Nutrition Research Center, Grand Forks, North Dakota, United States

REFERENCES:
- [Background] Roughead ZK, Johnson LK, Lykken GI, Hunt JR. Controlled high meat diets do not affect calcium retention or indices of bone status in healthy postmenopausal women. J Nutr. 2003 Apr;133(4):1020-6. doi: 10.1093/jn/133.4.1020. PMID 12672913
- [Derived] Cao JJ, Johnson LK, Hunt JR. A diet high in meat protein and potential renal acid load increases fractional calcium absorption and urinary calcium excretion without affecting markers of bone resorption or formation in postmenopausal women. J Nutr. 2011 Mar;141(3):391-7. doi: 10.3945/jn.110.129361. Epub 2011 Jan 19. PMID 21248199

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the Grand Forks, North Dakota community in November and December, 2007.
Pre-assignment Details: Of the 128 women who applied for the study, 56 did not meet the criteria, 46 declined, 4 were alternates, and 22 joined the study.
Groups:
- High Meat & High Potential Renal Acid Load - First: High meat and high potential renal acid load (high PRAL) diet followed by low meat and low potential renal acid load (low PRAL) diet.
- Low Meat & Low Potential Renal Acid Load - First: Low meat and low potential renal acid load (low PRAL) followed by High meat and high potential renal acid load (high PRAL) diet.
Period: Period: First Intervention
Arm/Group | High Meat & High Potential Renal Acid Load - First | Low Meat & Low Potential Renal Acid Load - First
Started | 10 | 12
Completed | 10 | 7
Not Completed | 0 | 5
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Protocol Violation | 0 | 3
Period: Period: Washout Period of 1 Week
Arm/Group | High Meat & High Potential Renal Acid Load - First | Low Meat & Low Potential Renal Acid Load - First
Started | 10 | 7
Completed | 10 | 7
Not Completed | 0 | 0
Period: Period: Second Intervention
Arm/Group | High Meat & High Potential Renal Acid Load - First | Low Meat & Low Potential Renal Acid Load - First
Started | 10 | 7
Completed | 9 | 7
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: Dietary Intervention: Crossover design, High meat and high potential renal acid load (high PRAL) diet and low meat and low potential renal acid load (low PRAL) diet, consumed in random order.
Arm/Group | Entire Study Population
Number analyzed (Participants) | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.9 (3.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Calcium Absorption
Description: After 3 weeks equilibration to the diet, the 2-day menu was extrinsically labeled with Calcium-47 radiotracer and retention was monitored for 28 days by whole body scintillation counting. Percent Calcium-47 absorbed was estimated from the y-intercept of the linear portion of a semilogarithmic plot of percent Calcium-47 retained vs time.
Time Frame: 18 weeks
Population: Analysis included only the 16 volunteers that completed both dietary interventions.
Measure: Mean (Standard Error); unit: percentage of Calcium-47 absorbed
Groups:
- High Meat - High Potential Renal Acid Load: High meat and high potential renal acid load (high PRAL) diet in either the first or second intervention period
- Low Meat - Low Potential Renal Acid Load: Low meat and low potential renal acid load (low PRAL) diet in either the first or second intervention period
Arm/Group | High Meat - High Potential Renal Acid Load | Low Meat - Low Potential Renal Acid Load
Number analyzed (Participants) | 16 | 16
percentage of Calcium-47 absorbed | 30.4 (2.4) | 25.4 (2.4)
Statistical Analysis 1: Comparison: High Meat - High Potential Renal Acid Load vs Low Meat - Low Potential Renal Acid Load; 16 subjects required to detect a difference in Calcium 47 absorption of 2 percentage points with 90% power, alpha = 0.05; Test type: Superiority or Other; p = 0.02, Mixed Models Analysis; Mixed model analysis of variance tested for treatment and feeding sequence effects; Mean Difference (Final Values) = 5, Standard Error of Mean 2

ADVERSE EVENTS:
Arm/Group | High Meat & High Potential Renal Acid Load - First | Low Meat & Low Potential Renal Acid Load - First
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/19
Other Adverse Events (participants affected / at risk) | 0/20 | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes